CLINICAL TRIAL: NCT04882917
Title: A First-in-human, Phase I, Open-label Study of the ATM Inhibitor M4076 in Participants With Advanced Solid Tumors (DDRiver Solid Tumors 410)
Brief Title: First-in-human Study of M4076 in Advanced Solid Tumors (DDRiver Solid Tumors 410)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: EMD Serono Research & Development Institute, Inc. (Industry)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Organization: EMD Serono (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MS201512_0010
Record Dates: First submitted 2021-05-07; First posted 2021-05-12 (Actual); Results first posted 2025-03-07 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Advanced Solid Tumors
Keywords: M4076; Maximum tolerated dose; Pharmacokinetics; Pharmacodynamics

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part 1A Dose Escalation: M4076 100 mg (Experimental): Participants received M4076 film coated tablets at a dose of 100 milligrams (mg), orally once daily in 21-day cycles, starting from Day 1 of each cycle disease progression, death, AE leading to discontinuation of study intervention(s), or withdrawal of consent, whichever occurred first, or End of Study
  Interventions: Drug: M4076
- Part 1A Dose Escalation: M4076 200 mg (Experimental): Participants received M4076 film coated tablets at a dose of 200 mg, orally once daily in 21-day cycles, starting from Day 1 of each cycle disease progression, death, AE leading to discontinuation of study intervention(s), or withdrawal of consent, whichever occurred first, or End of Study.
  Interventions: Drug: M4076
- Part 1A Dose Escalation: M4076 300 mg (Experimental): Participants received M4076 film coated tablets at a dose of 300 mg, orally once daily in 21-day cycles, starting from Day 1 of each cycle disease progression, death, AE leading to discontinuation of study intervention(s), or withdrawal of consent, whichever occurred first, or End of Study.
  Interventions: Drug: M4076
- Part 1A Dose Escalation: M4076 400 mg (Experimental): Participants received M4076 film coated tablets at a dose of 400 mg, orally once daily in 21-day cycles, starting from Day 1 of each cycle disease progression, death, AE leading to discontinuation of study intervention(s), or withdrawal of consent, whichever occurred first, or End of Study.
  Interventions: Drug: M4076

INTERVENTIONS:
Drug: M4076 — M4076 was administered orally.

SUMMARY:
The purpose of this study was to determine the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD), maximum tolerated dose (MTD) (if reached) and early signs of efficacy of M4076 monotherapy in participants with solid tumors in dose escalation (Part 1A). Once the recommended dose for expansion (RDE) was declared in Part 1A, a preliminary food effect cohort, Part 1B, will follow at the RDE determined from Part 1A.

ELIGIBILITY:
Inclusion Criteria:

* Participants with advanced solid tumors, for whom no standard of care therapy exists or for whom is not considered sufficiently effective, or who cannot tolerate standard of care
* Participants with Eastern Cooperative Oncology Group Performance status 0 or 1
* Adequate hematological, hepatic, and renal function as defined in the protocol
* Participants in Part 1B (the preliminary food effect assessment) must agree to provide paired tumor biopsies if not contraindicated for medical reasons
* Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* Clinically significant (i.e., active) uncontrolled intercurrent illness including, but not limited to:

  1. Active infection (i.e., requiring systemic antibiotics or antifungals)
  2. Uncontrolled arterial hypertension
  3. Severe cardiac arrhythmia requiring medication
  4. Cerebral vascular accident/stroke
* Has known ataxia telangiectasia
* Participants with tumors harboring previously identified ATM mutations
* Participants with hypersensitivity to the active substance or to any of the excipients of M4076
* Other protocol defined exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2021-05-24 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany
Locations (3):
- United States (2):
  - MD Anderson Center, Houston, Texas
  - NEXT Oncology, San Antonio, Texas
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
We are committed to enhancing public health through responsible sharing of clinical trial data. Following approval of a new product or a new indication for an approved product in both the US and the European Union, the study sponsor and/or its affiliated companies will share study protocols, anonymized patient data and study level data, and redacted clinical study reports with qualified scientific and medical researchers, upon request, as necessary for conducting legitimate research. Further information on how to request data can be found on our website http://bit.ly/IPD21

REFERENCES:
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=MS201512_0010
- See also: US Medical Information website, Medical Resources — https://medical.emdserono.com/en_US/home.html
- See also: DDRiver website — http://www.DDRiver-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 31 participants were screened, of which 22 participants received the study drug.
Pre-assignment Details: This study was to be conducted in 2 parts; Part 1A was the dose escalation phase and Part 1B was the expansion phase. However, the sponsor decided not to conduct the expansion phase (Part 2).
Period: Overall Study
Arm/Group | Part 1A Dose Escalation: M4076 100 mg | Part 1A Dose Escalation: M4076 200 mg | Part 1A Dose Escalation: M4076 300 mg | Part 1A Dose Escalation: M4076 400 mg
Started | 2 | 7 | 9 | 4
Completed | 0 | 6 | 5 | 1
Not Completed | 2 | 1 | 4 | 3
Not completed — Adverse Event | 0 | 1 | 2 | 2
Not completed — Withdrawal by Subject | 1 | 0 | 2 | 1
Not completed — COVID-19-related and COVID-19-non-related | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1A Dose Escalation: M4076 100 mg | Part 1A Dose Escalation: M4076 200 mg | Part 1A Dose Escalation: M4076 300 mg | Part 1A Dose Escalation: M4076 400 mg | Total
Number analyzed (Participants) | 2 | 7 | 9 | 4 | 22
Age, Continuous [Mean (Standard Deviation); unit: Years] | 74 (6.4) | 53 (7.0) | 60 (7.9) | 57 (5.7) | 58 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 5 | 4 | 3 | 13
  Male | 1 | 2 | 5 | 1 | 9
Race/Ethnicity, Customized [Number; unit: Participants]
  Ethnicity-Hispanic or Latino | 1 | 2 | 1 | 0 | 4
  Ethnicity-Not Hispanic or Latino | 1 | 5 | 8 | 4 | 18
  Race-Asian | 0 | 0 | 1 | 1 | 2
  Race-Black or African American | 0 | 0 | 1 | 0 | 1
  Race-Other | 0 | 2 | 0 | 0 | 2
  Race-White | 2 | 5 | 7 | 3 | 17

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experienced Dose Limiting Toxicities (DLTs) Assessed Using National Cancer Institute (NCI) Common Toxicity Criteria for Adverse Events (CTCAE) Version 5.0
Description: A DLT was defined as the occurrence of any of following events that were judged by the study investigator, received at least 80% of the planned cumulative dose during the DLT period of each study intervention and completed the DLT period or additionally, participants who did not receive 80% of the planned total dose of study intervention, but at least 80% dosing of a different dose cohort and finished the DLT period are eligible for the DLT analysis set to be analyzed in the highest dose cohort for which they received 80% of dosing.
Time Frame: Day 1 to Day 21 of Cycle 1 (21-day cycle)
Population: Dose escalation set included all participants who received at least 80 percent (%) of the planned cumulative dose during the DLT period (Period 1) and have completed the DLT Period or experienced at least one DLT during the DLT period, regardless of administered number of doses of study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1A Dose Escalation: M4076 100 mg | Part 1A Dose Escalation: M4076 200 mg | Part 1A Dose Escalation: M4076 300 mg | Part 1A Dose Escalation: M4076 400 mg
Number analyzed (Participants) | 2 | 5 | 7 | 4
Participants | 0 | 1 | 1 | 2

2. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Treatment Related TEAEs
Description: An Adverse event (AE) was defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease associated with the use of study drug, whether or not considered related to the study drug or worsening of pre-existing medical condition, whether or not related to study drug. A serious adverse event (SAE) was an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. The term TEAE is defined as AEs starting or worsening after the first intake of the study drug. TEAEs include both Serious TEAEs and non-serious TEAEs.
Time Frame: From the first dose of study drug administration until 30 days after the last dose of study drug administration (up to 603 days)
Population: Safety analysis set included all participants who were administered at least one dose of any study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1A Dose Escalation: M4076 100 mg | Part 1A Dose Escalation: M4076 200 mg | Part 1A Dose Escalation: M4076 300 mg | Part 1A Dose Escalation: M4076 400 mg
Number analyzed (Participants) | 2 | 7 | 9 | 4
Participants
  TEAEs | 2 | 7 | 9 | 4
  Treatment Related TEAEs | 1 | 2 | 8 | 4

3. Primary Outcome: Number of Participants With Clinically Significant Changes From Baseline in Vital Signs
Description: Vital sign assessments included assessments of heart rate, diastolic blood pressure, systolic blood pressure, weight, respiratory rate and temperature. Clinical significance was assessed by the investigator. Number of participants who with clinically significant changes from baseline in vital signs were reported.
Time Frame: Baseline (Day 1) up to 30 days after the last dose of study drug administration (up to 603 days)
Population: Safety analysis set included all participants who were administered at least one dose of any study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1A Dose Escalation: M4076 100 mg | Part 1A Dose Escalation: M4076 200 mg | Part 1A Dose Escalation: M4076 300 mg | Part 1A Dose Escalation: M4076 400 mg
Number analyzed (Participants) | 2 | 7 | 9 | 4
Participants | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Change From Baseline in Laboratory Test Abnormalities to Grade 3 or Higher Severity Based on NCI-CTCAE Version 5.0
Description: The laboratory measurements included hematology and biochemistry values were graded with National Cancer Institute - Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0 toxicity grades (where Grade 1 = mild, Grade 2 = moderate, Grade 3 = severe, Grade 4 = life threatening and Grade 5 = death). Number of participants with change from baseline to grade 3 or higher values for the hematology and biochemistry were reported.
Time Frame: Baseline (Day 1) up to 30 days after the last dose of study drug administration (up to 603 days)
Population: Safety analysis set included all participants who were administered at least one dose of any study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1A Dose Escalation: M4076 100 mg | Part 1A Dose Escalation: M4076 200 mg | Part 1A Dose Escalation: M4076 300 mg | Part 1A Dose Escalation: M4076 400 mg
Number analyzed (Participants) | 2 | 7 | 9 | 4
Participants
  Grade>=3 Alanine Aminotransferase High | 0 | 0 | 0 | 1
  Grade>=3 Aspartate Aminotransferase High | 0 | 0 | 0 | 1
  Grade>=3 Alkaline Phosphatase High | 0 | 0 | 0 | 1
  Grade>=3 Gamma Glutamyl Transferase High | 0 | 0 | 0 | 1
  Grade>=3 Bilirubin High | 0 | 1 | 0 | 0
  Grade>=3 Lipase High | 0 | 1 | 0 | 0
  Grade>=3 Sodium Low | 0 | 0 | 1 | 0
  Grade>=3 Potassium High | 0 | 1 | 0 | 0
  Grade>=3 Potassium Low | 0 | 1 | 0 | 0
  Grade>=3 Calcium High | 0 | 1 | 0 | 0
  Grade>=3 Hemoglobin Low | 0 | 1 | 2 | 1
  Grade>=3 Lymphocytes Low | 0 | 3 | 3 | 2

5. Primary Outcome: Number of Participants With Clinically Significant Changes From Baseline in Electrocardiogram (ECG) Values
Description: ECG parameters included rhythm, heart rate (as measured by RR interval), PR interval, QRS duration, QT intervals, and corrected QT(QTc) intervals. Clinical significance was determined by the investigator. Number of participants with clinically significant change from baseline in 12-lead ECG were reported.
Time Frame: Baseline (Day 1) up to 30 days after the last dose of study drug administration (up to 603 days)
Population: Safety analysis set included all participants who were administered at least one dose of any study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1A Dose Escalation: M4076 100 mg | Part 1A Dose Escalation: M4076 200 mg | Part 1A Dose Escalation: M4076 300 mg | Part 1A Dose Escalation: M4076 400 mg
Number analyzed (Participants) | 2 | 7 | 9 | 4
Participants | 0 | 0 | 0 | 0

6. Secondary Outcome: Number of Participants With Confirmed Objective Response According to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) as Assessed by Investigator
Description: Confirmed objective response was defined as the number of participants with a confirmed objective response of complete response (CR) or partial response (PR). CR: Disappearance of all evidence of target and non-target lesions. PR: At least 30% reduction from baseline in the sum of the longest diameter (SLD) of all lesions. Confirmed CR = at least 2 determinations of CR at least 4 weeks apart and before progression. Confirmed PR = at least 2 determinations of PR at least 4 weeks apart and before progression (and not qualifying for a CR).
Time Frame: Time from first study treatment up to 603 days
Population: Full analysis set included all participants who were administered at least one dose of any study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1A Dose Escalation: M4076 100 mg | Part 1A Dose Escalation: M4076 200 mg | Part 1A Dose Escalation: M4076 300 mg | Part 1A Dose Escalation: M4076 400 mg
Number analyzed (Participants) | 2 | 7 | 9 | 4
Participants | 0 [0.00 to 84.19] | 0 [0.00 to 40.96] | 0 [0.00 to 33.63] | 0 [0 to 15.44]

7. Secondary Outcome: Duration of Response (DOR) According to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) as Assessed by Investigator
Description: DOR was defined for participants with confirmed response, as the time from first documentation of objective response (Complete Response [CR] or Partial Response [PR]) to the date of first documentation of progression disease (PD) or death due to any cause, whichever occurred first. CR: Disappearance of all evidence of target and non-target lesions. PR: At least 30% reduction from baseline in the SLD of all lesions. PD: At least a 20 percent (%) increase in the SLD, taking as reference the smallest SLD recorded from baseline or the appearance of 1 or more new lesions.
Time Frame: Time from first documentation of objective response to the date of first documentation of PD or death due to any cause, assessed up to 603 days
Population: None of the participants showed objective response.
Arm/Group | Part 1A Dose Escalation: M4076 100 mg | Part 1A Dose Escalation: M4076 200 mg | Part 1A Dose Escalation: M4076 300 mg | Part 1A Dose Escalation: M4076 400 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0

8. Secondary Outcome: Progression-Free Survival (PFS) According to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) Assessed by Investigators
Description: PFS is defined as the time (in months) from date of first administration of study intervention to the date of the first documentation of progressive disease (PD) or death due to any cause, whichever occurs first. PD is defined as at least a 20 percent (%) increase in the sum of the longest diameter (SLD), taking as reference the smallest SLD recorded from baseline or the appearance of 1 or more new lesions. PFS was to be estimated using Kaplan-Meier (KM) plots.
Time Frame: Time from the first dose of study intervention until occurrence of PD, death due to any cause or last tumor assessment (assessed up to 603 days)
Population: Full analysis set included all participants who were administered at least one dose of any study intervention.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part 1A Dose Escalation: M4076 100 mg | Part 1A Dose Escalation: M4076 200 mg | Part 1A Dose Escalation: M4076 300 mg | Part 1A Dose Escalation: M4076 400 mg
Number analyzed (Participants) | 2 | 7 | 9 | 4
months | NA [NA to NA] — Median (and corresponding 95% CI) could not be estimated by KM estimates as there was no event of interest. | 1.1 [0.20 to 1.58] | 1.3 [0.69 to 2.60] | NA [1.22 to NA] — Median (and corresponding 95% CI) could not be estimated due to low number of events of interest (1 participant).

9. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to Last Sampling Time (AUClast) of M4076
Description: Area under the plasma concentration vs time curve from time zero to the last sampling time t at which the concentration was at or above the lower limit of quantification (LLOQ). AUC0-tlast was to be calculated according to the mixed log-linear trapezoidal rule.
Time Frame: Day 1 and Day 8
Population: Pharmacokinetic Analysis Set included all participants who were administered at least one dose of study intervention. Here, "Number analyzed" signifies those participants who were evaluable for this outcome measure at specified timepoints.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*nanograms per milliliter
Arm/Group | Part 1A Dose Escalation: M4076 100 mg | Part 1A Dose Escalation: M4076 200 mg | Part 1A Dose Escalation: M4076 300 mg | Part 1A Dose Escalation: M4076 400 mg
Number analyzed (Participants) | 2 | 7 | 9 | 4
hour*nanograms per milliliter
  Day 1 | NA (NA) — Based on pre-specified criteria, statistical analysis was only performed if more than 2 participants have reportable parameter values. | 37000 (34.1) | 50500 (45.1) | 76600 (44.3)
  Day 8: number analyzed (Participants) | 2 | 5 | 8 | 3
  Day 8 | NA (NA) — Based on pre-specified criteria, statistical analysis was only performed if more than 2 participants have reportable parameter values. | 36500 (109.2) | 56500 (67.6) | 85900 (40.8)

10. Secondary Outcome: Area Under Plasma Concentration-Time Curve From Time Zero Extrapolated to Infinity (AUC0-inf) of M4076
Description: The AUC from time zero (dosing time) extrapolated to infinity, based on the predicted value for the concentration at tlast, as estimated using the linear regression from lambda z determination. AUC0-inf = AUC0-tlast +Clast pred/ lambda z (single dose only)
Time Frame: Day 1 and Day 8
Population: Pharmacokinetic Analysis Set included all participants who were administered at least one dose of study intervention. Here, "Number of participants analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Part 1A Dose Escalation: M4076 100 mg | Part 1A Dose Escalation: M4076 200 mg | Part 1A Dose Escalation: M4076 300 mg | Part 1A Dose Escalation: M4076 400 mg
Number analyzed (Participants) | 2 | 6 | 6 | 3
h*ng/mL
  Day 1 | NA (NA) — Based on pre-specified criteria, statistical analysis was only performed if more than 2 participants have reportable parameter values. | 39200 (40.3) | 44900 (49.9) | 69800 (20.4)
  Day 8: number analyzed (Participants) | 0 | 0 | 0 | 0

11. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of M4076
Description: Cmax was obtained directly from the concentration versus time curve.
Time Frame: Day 1 and Day 8
Population: Pharmacokinetic Analysis Set included all participants who were administered at least one dose of study intervention, have no clinically important protocol deviations or important events affecting pharmacodynamics, and provide the baseline and at least one measurable pharmacodynamics endpoint post dose. Here, "Number of participants analyzed" signifies those participants who were evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Part 1A Dose Escalation: M4076 100 mg | Part 1A Dose Escalation: M4076 200 mg | Part 1A Dose Escalation: M4076 300 mg | Part 1A Dose Escalation: M4076 400 mg
Number analyzed (Participants) | 2 | 6 | 8 | 3
nanogram per milliliter (ng/mL)
  Day 1: number analyzed (Participants) | 2 | 6 | 6 | 3
  Day 1 | NA (NA) — Based on pre-specified criteria, statistical analysis was only performed if more than 2 participants have reportable parameter values | 4080 (26.5) | 6270 (20.3) | 8510 (30.1)
  Day 8: number analyzed (Participants) | 2 | 5 | 8 | 3
  Day 8 | NA (NA) — Based on pre-specified criteria, statistical analysis was only performed if more than 2 participants have reportable parameter values. | 4690 (52.5) | 6730 (26.3) | 9600 (22.8)

12. Secondary Outcome: Absolute Changes From Baseline in Ataxia-Telangiectasia Mutated (ATM) Pathway Readouts Assessed by Flow Cytometry and Immunohistochemistry: p-ATM
Description: Phosphorylated ataxia-telangiectasia mutated (p-ATM) is measured by flow cytometry and immunohistochemistry. Absolute change from baseline was to be reported.
Time Frame: Baseline up to Day 23
Population: Data for p-ATM was not generated due to insufficient samples as all Peripheral Blood Mononuclear Cells (PBMC) samples were exhausted in gamma-H2AX analysis. Hence no data was collected.
Arm/Group | Part 1A Dose Escalation: M4076 100 mg | Part 1A Dose Escalation: M4076 200 mg | Part 1A Dose Escalation: M4076 300 mg | Part 1A Dose Escalation: M4076 400 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0

13. Secondary Outcome: Absolute Changes From Baseline in Ataxia-Telangiectasia Mutated (ATM) Pathway Readouts Assessed by Flow Cytometry and Immunohistochemistry: p-CHK2
Description: p-CHK2 is measured by flow cytometry and immunohistochemistry. Absolute change from baseline was to be reported.
Time Frame: Baseline up to Day 23
Population: Data for p-CHK2 was not generated as no fresh tumor biopsies were collected. Hence no data was collected.
Arm/Group | Part 1A Dose Escalation: M4076 100 mg | Part 1A Dose Escalation: M4076 200 mg | Part 1A Dose Escalation: M4076 300 mg | Part 1A Dose Escalation: M4076 400 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0

14. Secondary Outcome: Relative Changes From Baseline in Ataxia-Telangiectasia Mutated (ATM) Pathway Readouts Assessed by Flow Cytometry and Immunohistochemistry: p-ATM
Description: Phosphorylated ataxia-telangiectasia mutated (p-ATM) is measured by flow cytometry and immunohistochemistry. Relative change from baseline was to be reported.
Time Frame: Baseline up to Day 23
Population: as for outcome 12
Arm/Group | Part 1A Dose Escalation: M4076 100 mg | Part 1A Dose Escalation: M4076 200 mg | Part 1A Dose Escalation: M4076 300 mg | Part 1A Dose Escalation: M4076 400 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0

15. Secondary Outcome: Relative Changes From Baseline in Ataxia-Telangiectasia Mutated (ATM) Pathway Readouts Assessed by Flow Cytometry and Immunohistochemistry: p-CHK2
Description: p-CHK2 is measured by flow cytometry and immunohistochemistry. Relative change from baseline was to be reported.
Time Frame: Baseline up to Day 23
Population: Data for p-CHK2 was not generated as no fresh tumor biopsies were collected. Hence no data was collected.
Arm/Group | Part 1A Dose Escalation: M4076 100 mg | Part 1A Dose Escalation: M4076 200 mg | Part 1A Dose Escalation: M4076 300 mg | Part 1A Dose Escalation: M4076 400 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0

16. Secondary Outcome: Absolute Values in Ataxia-Telangiectasia Mutated (ATM) Pathway Readouts Assessed by Flow Cytometry and Immunohistochemistry: Gamma-H2AX
Description: gamma-H2AX is measured by flow cytometry and immunohistochemistry. Absolute values were reported for each participant as descriptive data for this outcome measure was not calculated. P= Part, D=Day, H=Hour in the below mentioned categories. Mean Fluorescent Intensity (MFI) is a number generated by the flow cytometer; an instrument that measures the fluorescent signal emitted by a sample. The stronger the fluorescent signal, the higher the MFI value detected by the instrument's acquisition software. The values displayed in the system represent each MFI measurement at different time points, with the MFI value for the blank sample subtracted.
Time Frame: Baseline up to Day 23
Population: The pharmacodynamics (Pd) Analysis Set consisted of all participants, who received at least one dose of study intervention, had no clinically important protocol deviations or important events affecting Pd, and provide the baseline and at least one measurable Pd endpoint postdose. Participants will be analyzed per the actual study intervention they received.
Measure: Number; unit: Mean fluorescence intensity
Groups:
- Part 1A Dose Escalation: M4076 mg (All Participants): Participants received M4076 film coated tablets at a dose of 100, 200, 300 or 400 milligrams (mg), orally once daily in 21-day cycles, starting from Day 1 of each cycle disease progression, death, AE leading to discontinuation of study intervention(s), or withdrawal of consent, whichever occurred first, or End of Study
Arm/Group | Part 1A Dose Escalation: M4076 mg (All Participants)
Number analyzed (Participants) | 21
Mean fluorescence intensity
  Participant1(P1AD1-2H Postdose) | 1316
  Participant1(P1AD1-4H Postdose) | 1037
  Participant1(P1AD1-6H Postdose) | 3127
  Participant1(P1AD1-Predose) | 1612
  Participant1(P1AD2-2-4H Postdose) | 347
  Participant1(P1AD2-Predose) | 1925
  Participant1(P1A/1BD22-2H Postdose | 1030
  Participant1(P1A/1BD22-4H Postdose) | 1023
  Participant1(P1A/1BD22-Predose) | 1461
  Participant2(P1AD1-6H Postdose) | 896
  Participant2(P1AD2-2-4H Postdose) | 143
  Participant2(P1A/1BD22-2H Postdose) | 753
  Participant2(P1A/1BD22-Predose) | 1441
  Participant3(P1AD1-2H Postdose) | 5555
  Participant3(P1AD1-4H Postdose) | 4432
  Participant3(P1AD2-2H-4H Postdose) | 1504
  Participant3(P1AD2-4H Predose) | 2649
  Participant4(P1AD1-2H Postdose) | 879
  Participant4(P1AD1-4H Potdose) | 395
  Participant4(P1AD1-6H Postdose) | 702
  Participant4(P1AD1-Predose) | -34
  Participant4(P1AD2-2H-4H Postdose) | 1045
  Participant4(P1AD2-Predose) | 1057
  Participant5(P1AD1-2H Postdose) | 195
  Participant5(P1AD1-4H Postdose) | 171
  Participant5(P1AD1-6H Postdose) | 75
  Participant5(P1AD1-Predose) | 144
  Participant5(P1AD2-2H-4H Postdose) | 0
  Participant5(P1AD2-Predose) | 22
  Participant6(P1AD1-2H Postdose) | 57
  Participant6(P1AD1-4H Postdose) | 138
  Participant6(P1AD1-6H Postdose) | 116
  Participant6(P1AD1-4H Predose) | 206
  Participant6(P1AD2-2H-4H Postdose) | 1
  Participant6(P1AD2- Predose) | 29
  Participant6(P1A/1BD22-2H Postdose) | 994
  Participant6(P1A/1BD22-4H Postdose) | 786
  Participant6(P1A/1BD22-Predose) | 2371
  Participant7(P1A/1BD22-4H Postdose) | 5397
  Participant7(P1A/1BD22-2H-4H Postdose) | 770
  Participant7(P1AD2-Predose) | 1103
  Participant8(P1AD1-2H Postdose) | 1775
  Participant8(P1AD1-4H Postdose) | 1504
  Participant8(P1AD1-6H Postdose) | 854
  Participant8(P1AD1-Predose) | 2294
  Participant8(P1AD1-2H-4H Postdose) | 381
  Participant8(Part1AD2-Predose) | 910
  Participant9(P1AD1-2H Postdose) | 2836
  Participant9(P1AD1-4H Postdose) | 1499
  Participant9(P1AD1-6H Postdose) | 1901
  Participant9(P1AD1-Predose) | -4092
  Participant9(P1AD2-2H-4H Postdose) | 2392
  Participant9(P1A/1BD22-2H Postdose) | 2795
  Participant9(P1A/1BD22-4H Postdose) | 3375
  Participant9(P1A/1BD22-Predose) | 3412
  Participant10(P1A/1BD22-2H Postdose) | 747
  Participant10(P1A/1BD22-4H Postdose) | 1186
  Participant10(P1A/1BD22-Predose) | 1608
  Participant10(P1AD1-2H Postdose) | 2014
  Participant10(P1AD1-4H Postdose) | 1522
  Participant10(P1AD1-2H-4H Postdose) | 2363
  Participant10(P1AD2-Predose) | 1018
  Participant11(P1AD1-2H Postdose) | 2432
  Participant11(P1AD1-4H Postdose) | 1282
  Participant11(P1A/1BD22-2H Postdose) | -802
  Participant11(P1A/1BD22- Predose) | -904
  Participant11(P1A/1BD22-4H Postdose) | -1708
  Participant12(P1AD1-2H Postdose) | 3613
  Participant12(P1AD1-Predose) | 5007
  Participant12(P1AD2-2H-4H Postdose) | 4438
  Participant12(P1AD2-Predose) | 4088
  Participant13(P1AD2-2H-4H Postdose) | 2650
  Participant13(P1AD2-Predose) | 2342
  Participant13(P1A/1BD22-2H Postdose) | 1194
  Participant13(P1A/1BD22-4H Postdose) | -70
  Participant13(P1A/1BD22 Predose) | 2532
  Participant14(P1AD1-2H Postdose) | 329
  Participant14(P1AD1-4H Postdose) | 139
  Participant14(P1AD1-6H Postdose) | 194
  Participant14(P1AD1-Predose) | 704
  Participant14(P1AD2-2H-4H Postdose) | 208
  Participant14(P1AD2-Predose) | 115
  Participant14(P1A/1BD22-Predose) | 210
  Participant15(P1AD1-2H Postdose) | 829
  Participant15(P1AD1-4H Postdose) | 1006
  Participant15(P1AD1-6H Postdose) | 596
  Participant15(P1AD1-Predose) | 1808
  Participant15(P1AD2-2H-4H Postdose) | 1742
  Participant15(P1AD2-2H Predose) | 2074
  Participant16(P1AD1-2H Postdose) | 562
  Participant16(P1AD1-4H Postdose) | 416
  Participant16(P1AD1-6H Postdose) | 554
  Participant16(P1AD1-Predose) | 644
  Participant16(P1AD2-2H-4H Postdose) | 704
  Participant17(P1AD1-2H Postdose) | 2200
  Participant17(P1AD1-4H Postdose) | 799
  Participant17(P1AD2-2H-4H Postdose) | 729
  Participant17(P1AD2-Predose) | 3157
  Participant18(P1AD1-6H Postdose) | 845
  Participant18(P1AD1-Presdose) | 1261
  Participant18(P1AD2-2H-4H Postdose) | 2257
  Participant19(P1AD1-2H Postdose) | 2182
  Participant19(P1AD1-4H Postdose) | 1831
  Participant19(P1AD1-6H Postdose) | 1871
  Participant19(P1AD1-Predose) | -2466
  Participant19(P1AD2-2H-4H Postdose) | 1677
  Participant19(P1AD2-Predose) | 4862
  Participant20(P1A/1BD22-2H Postdose) | 11119
  Participant20(P1AD1-2H Postdose | 1967
  Participant20(P1AD1-4H Postdose | -593
  Participant20(P1AD1-6H Postdose | 2977
  Participant20(P1AD1-Predose) | 262
  Participant20(P1AD2-2H-4H Postdose) | 1860
  Participant20(P1AD2-Predose) | 3150
  Participant21(P1AD1-2H Postdose) | 660
  Participant21(P1AD1-4H Postdose) | 1392
  Participant21(P1AD1-6H Postdose) | 787
  Participant21(P1AD1 Predose) | 2280
  Participant21(P1AD2-2H-4H Postdose) | -128
  Participant21(P1AD2 Predose) | 1389

ADVERSE EVENTS:
Time Frame: Up to 603 days
Arm/Group | Part 1A Dose Escalation: M4076 100 mg | Part 1A Dose Escalation: M4076 200 mg | Part 1A Dose Escalation: M4076 300 mg | Part 1A Dose Escalation: M4076 400 mg
All-Cause Mortality (participants affected / at risk) | 0/2 | 4/7 | 1/9 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/2 | 4/7 | 2/9 | 3/4
Other Adverse Events (participants affected / at risk) | 2/2 | 7/7 | 9/9 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1A Dose Escalation: M4076 100 mg (N=2) | Part 1A Dose Escalation: M4076 200 mg (N=7) | Part 1A Dose Escalation: M4076 300 mg (N=9) | Part 1A Dose Escalation: M4076 400 mg (N=4)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Immune system disorder (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Liver abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spontaneous bacterial peritonitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary tract stoma complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1A Dose Escalation: M4076 100 mg (N=2) | Part 1A Dose Escalation: M4076 200 mg (N=7) | Part 1A Dose Escalation: M4076 300 mg (N=9) | Part 1A Dose Escalation: M4076 400 mg (N=4)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Eye irritation (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 3 (3) | 1 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Fatigue (General disorders) | 0 (0) | 2 (2) | 4 (4) | 3 (3)
Gait disturbance (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 2 (3) | 4 (4) | 2 (3)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Liver abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Spontaneous bacterial peritonitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 2 (3) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 2 (2) | 1 (3) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 1 (1) | 2 (2) | 3 (4)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
White blood cell count increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-10-27): https://cdn.clinicaltrials.gov/large-docs/17/NCT04882917/Prot_000.pdf
  • Statistical Analysis Plan (2022-12-19): https://cdn.clinicaltrials.gov/large-docs/17/NCT04882917/SAP_001.pdf